CLINICAL TRIAL: NCT01344707
Title: Open Label, Dose Escalation Study of 4SC-202 in Patients With Advanced Hematologic Malignancies: First-In-Man Study of a Newly Developed, Oral Histone Deacetylase Inhibitor
Brief Title: Oral Histone Deacetylase Inhibitor 4SC-202 in Patients With Advanced Hematologic Malignancies (TOPAS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: 4SC AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4SC-202-1-2010
Record Dates: First submitted 2011-04-12; First posted 2011-04-29 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2014-01

CONDITIONS: Advanced Hematologic Malignancies
Keywords: Hematologic Malignancies; Acute Myeloid Leukemia (AML); Acute Lymphocytic Leukemia (ALL); Chronic Lymphocytic Leukemia (CLL); Multiple Myeloma (MM); Myelodysplastic Syndrome (MDS); Malignant Lymphomas; Histone Deacetylase (HDAC); 4SC-202; Phase I
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma; Myelodysplastic Syndromes; Lymphoma | interventions — domatinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 4SC-202 — oral administration dose escalation twice daily (bid)or three times a day (tid) continuous dosing for 21 days per cycle

SUMMARY:
The purpose of this study is to determine the Maximum Tolerated Dose, Dose Limiting Toxicities and optimal dosing schedule of 4SC-202 investigating its safety, tolerability and pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, age ≥ 18 years.
* Patients with Acute Myeloid Leukemia (AML), Acute Lymphocytic Leukemia (ALL), Chronic Lymphocytic Leukemia (CLL), Multiple Myeloma (MM),Myelodysplastic Syndrome (MDS) or malignant lymphoma which are relapsed and/or refractory to standard therapy or for which no standard therapy exists. Patients who are not eligible for curative stem cell transplantation or patients who have refused or are not eligible for frontline (chemo-) therapy may also be included.
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2.
* Patients must have a live expectancy of 12 weeks or more.
* Patients must have adequate bone marrow reserve as well as adequate renal and hepatic function and serum electrolytes within a clinically acceptable range.
* Patients must have recovered from any treatment-related toxicities (to Grade 0 or 1 according to Common Terminology Criteria for Adverse Events (CTCAE); except for alopecia, fatigue and Grade 1 neurotoxicity) prior to registration.

Exclusion Criteria:

* Patients who have received previous treatment with an HDAC inhibitor.
* Patients with any gastrointestinal disorder that could interfere with the absorption of 4SC-202
* Patients who are unable to take oral medication.
* Patients with a history of other malignancies unless having undergone definitive treatment more than 5 years prior to entry into the study and without evidence of recurrent malignant disease, excluding patients with basal cell carcinoma of the skin; superficial carcinoma of the bladder; carcinoma of the prostate with a current prostate specific antigen (PSA) value of < 0.1 ng/ml; or cervical intraepithelial neoplasia.
* Patients with a history of, who were treated for, or who are suspected of having, hepatitis B, hepatitis C or human immunodeficiency virus (HIV). Patients suspected of having any of these conditions should undergo appropriate evaluations prior to being enrolled in the study.
* Patients with precedent anti-cancer therapy including chemotherapy, radiotherapy, endocrine therapy, immunotherapy or use of other investigational agents within the last two weeks or a longer period depending on the known PK characteristics of the agents used.
* Patients with history or current evidence of clinically relevant allergies or idiosyncrasy to drugs (especially of similar chemical composition to the study drug) or food.
* Patients with symptomatic brain metastases/central nervous system (CNS) involvement.
* Patients with significant cardiovascular disease including unstable angina pectoris, uncontrolled hypertension, congestive heart failure (New York Heart Association (NYHA) Class III or IV) related to primary cardiac disease, a condition requiring anti-arrhythmic therapy, ischemic or severe valvular heart disease, or a myocardial infarction within 6 months prior to the trial entry.
* Patients with a marked baseline prolongation of QT/QTc interval, e.g., repeated demonstration of a QTc interval > 450 msec (Grade 1 CTCAE); Long-QT-Syndrome; the required use of concomitant medication on 4SC-202 dosing days that may cause Torsade de Pointes.
* Therapy with agents known to prolong the QT interval, such as certain antibiotics (i.e. erythromycin, clarithromycin), antidepressants (i.e. doxepin, amitryptilin) or neuroleptics (i.e. haloperidol, clozapin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2011-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Determination of Dose Limiting Toxicities of 4SC-202 | 6 weeks
Determination of Safety of 4SC-202 | 6 weeks
  The safety and tolerability will be determined by occurrence of adverse events (AEs), vital signs (VS) [body temperature, weight, blood pressure (BP), pulse rate], electrocardiogram (ECG), performance status and clinical laboratory parameters.
Determination of Pharmacokinetic Profile of 4SC-202 | 3 weeks
  The plasma concentrations of 4SC-202 will be determined at the following time-points:
  Cycle 1 Day 1: Pre-dose, 0.5 h, 1 h, 2 h, 3 h, 4 h, 5 h, 8 h, 24 h p.a. Cycle 1 Day 5: Pre-dose, 0.5 h, 1h, 2h Cycle 1 Day 14: Pre-dose, 0.5 h, 1 h, 2 h, 3 h, 4 h, 5 h, 8 h, 24 h p.a. Cycle 2 Day 1: Pre-dose, 0.5 h, 1 h, 2 h, 3 h, 4 h, 5 h, 8 h, 24 h p.a. using AUC0-infinity, AUClast, Cmax, tmax, t1/2, CL/F
Determination of Maximum Tolerated Dose of 4SC-202 | 6 weeks
Determination of Tolerability of 4SC-202 | 6 weeks
  The safety and tolerability will be determined by occurrence of adverse events (AEs), vital signs (VS) [body temperature, weight, blood pressure (BP), pulse rate], electrocardiogram (ECG), performance status and clinical laboratory parameters.

SECONDARY OUTCOMES:
Assessment of potential anticancer activity of 4SC-202 | 6 weeks
  The assessment will be performed by assessment of tumor response, duration of response and progression free survival
Histone deacetylase (HADAC) inhibition in peripheral mononuclear cells | 6 weeks
Histone acetylation in peripheral mononuclear cells | 6 weeks
Gene expression analysis in peripheral blood | 6 weeks
Cytokine and miRNA levels in plasma | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Engert, Prof. MD, Principal Investigator — Universitätsklinikum Köln
Locations (3):
- Germany (3):
  - Universiätsklinikum Köln, Cologne
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Universitätsklinikum Würzburg, Würzburg